CLINICAL TRIAL: NCT07335445
Title: Enhancing Screening Practices for Barrett's Esophagus
Brief Title: Enhancing Screening Practices for BE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Arvind Trindade, MD, FACG, FASGE, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2025000949
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Barrett's Esophagus
Keywords: screening; barrett's esophagus; barrett's
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- Intervention (Active Comparator)
  Interventions: Other: Screening Reminder

INTERVENTIONS:
Other: Screening Reminder — A reminder to screen this patient for Barrett's esophagus (BE) will be sent to the provider before the patient's scheduled appointment. The reminder will provide details about which criteria this patient meets in order to indicate that BE screening should be initiated.
  Arms: Intervention

SUMMARY:
Previous studies have shown that screening for Barrett's esophagus (BE), the main risk factor for esophageal adenocarcinoma, is under-utilized in the primary care setting. In fact less than 35% of eligible patients are screened despite endorsement for screening by the major GI societies in patients with risk factors. The purpose of this study is to examine current screening practices and determine if implementation of screening reminders can optimize screening practices for Barrett's Esophagus within a large, academic based healthcare system in NJ.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a pre-malignant mucosal transformation of the distal esophageal mucosal lining whereby the metaplastic columnar epithelium replaces squamous epithelium of the esophagus. BE is the main risk factor to develop esophageal adenocarcinoma. The etiology of BE is complex and likely multifactorial, with several factors including gastrointestinal reflux (GERD), genetic factors, environmental triggers, immunoregulatory defects playing a role. It is well known that the transformation of cells lining the distal esophagus is due to chronic repeated insults by longstanding GERD.

A significant proportion of patients diagnosed with BE are discovered during endoscopic evaluation of middle-aged and older adults however a majority of cases are unrecognized. The vast majority of patients (up to 90%) with EAC have never had a diagnosis of BE. A major limitation of BE screening are those individuals with silent or asymptomatic GERD. In a study evaluating the sensitivity of guidelines by determining the proportion of prevalent EAC that met screening criteria for BE by American College of Gastroenterology (ACG) or the British Society of Gastroenterology (BSG) guidelines, 54.9% of the US patients and 38.9% of the UK patients would not have been identified by current screening guidelines. Furthermore, the reason most patients (US, 86.5%; UK, 61.4%) did not meet screening guidelines was the lack of symptomatic GERD.

Currently, upper endoscopy with biopsies remains the gold standard for the diagnosis of BE however there is a significant need for other, non-invasive screening tools that are easy to implement, cost-friendly, and patient friendly. Other options include trans-nasal endoscopy and non-endoscopic cell collection devices which can be used in the outpatient setting and avoids need for sedation. Trans-nasal endoscopy remains costly, operator-dependent, and uncomfortable or distressing to patients. Current non-endoscopic cell collection devices include Cytosponge (Medtronic GI Solutions), EsoCheck (Lucid Diagnostics), and EsophaCap (Capnostics) which have demonstrated excellent safety, tolerability, and sensitivity for the diagnosis of BE. Nonendoscopic devices are currently an approved method of screening per the 2022 American College of Gastroenterology (ACG) society guidelines on diagnosis of BE.

The presence of metabolic disease increases the risk of developing cancer. Early studies suggested the presence of metabolic syndrome and visceral fat (eg, MASLD, pancreatic fatty infiltration) are associated with BE and typically portray higher risk for progression to dysplasia or neoplasia. Current standard is EGD for screening of BE and surveillance determined by histology and length of mucosal changes. The role of evaluation for visceral adiposity, either via cross-sectional imaging or endoscopic ultrasound, has not been elucidated. Factoring visceral adiposity may allow the investigators to risk-stratify patients for screening or optimize surveillance strategies to prevent progression to EAC.

This is a single center randomized controlled trial examining whether implementation of screening reminders for eligible patients will increase BE screening rates. The investigators will enroll 8 practices (see below) in the New Brunswick area. 4 practices will be randomized to the screening reminder arm and 4 practices will be randomized to the no reminder screening arm. In each arm baseline data will be collected on BE screening rates for the practice prior to the study for comparison.

The screening reminder arm will undergo the following. Patient's medical charts will be screened via epic to determine if patients meet criteria for BE screening per the ACG (American College of Gastroenterology) or ASGE (American Society of GI Endoscopy) guidelines. Charts will be screened by a gastroenterology fellow on the study team or a gastroenterology attending on the study team. If patients qualify for screening, the provider will receive an email and Epic chat the day before the patient's office appointment with the provider letting them know which patients on their panel qualify for screening for BE.

Providers in both arms of the study will be notified of GI services to help screen patients for BE prior the study inception, including referral to GI clinic for nonendoscopic screening.

BE screening is part of standard of care for patients who meet criteria, as defined by ACG/ASGE guidelines. Sending reminders to primary care offices/staff is not standard of care. The 8 practices are affiliated with RWJ Barnabas Health Medical group. Reminders (email or Epic chat) will be sent the day before the patient's scheduled appointment with the provider. Data regarding demographics, comorbidities, and presence of other factors that qualify patients into BE screening will be recorded. The investigators will then record which patients were or were not screened for BE with either invasive (eg, EGD) or non-invasive measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have a scheduled appointment with a participating provider

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
BE screening rate | 1 year
  Percentage increase in BE screening compared to each arm's historical control BE screening rate from the year prior.

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Trindade, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, following deidentification. Data will only be shared upon request, for an approved proposal, after review and approval by Rutgers University.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal, following approval by Rutgers University.

REFERENCES:
- [Background] Muthusamy VR, Wani S, Gyawali CP, Komanduri S; CGIT Barrett's Esophagus Consensus Conference Participants. AGA Clinical Practice Update on New Technology and Innovation for Surveillance and Screening in Barrett's Esophagus: Expert Review. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2696-2706.e1. doi: 10.1016/j.cgh.2022.06.003. Epub 2022 Jul 3. PMID 35788412
- [Background] Saha B, Vantanasiri K, Mohan BP, Goyal R, Garg N, Gerberi D, Kisiel JB, Singh S, Iyer PG. Prevalence of Barrett's Esophagus and Esophageal Adenocarcinoma With and Without Gastroesophageal Reflux: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2024 Jul;22(7):1381-1394.e7. doi: 10.1016/j.cgh.2023.10.006. Epub 2023 Oct 24. PMID 37879525
- [Background] Sawas T, Zamani SA, Killcoyne S, Dullea A, Wang KK, Iyer PG, Fitzgerald RC, Katzka DA. Limitations of Heartburn and Other Societies' Criteria in Barrett's Screening for Detecting De Novo Esophageal Adenocarcinoma. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1709-1718. doi: 10.1016/j.cgh.2021.10.039. Epub 2021 Oct 29. PMID 34757196
- [Background] Nguyen TH, Thrift AP, Rugge M, El-Serag HB. Prevalence of Barrett's esophagus and performance of societal screening guidelines in an unreferred primary care population of U.S. veterans. Gastrointest Endosc. 2021 Feb;93(2):409-419.e1. doi: 10.1016/j.gie.2020.06.032. Epub 2020 Jun 19. PMID 32565183